CLINICAL TRIAL: NCT01153503
Title: Ultrasound-guided Transversus Abdominis Plane Block After Abdominal Hysterectomy: a Prospective Randomized Controlled Trial
Brief Title: Ultrasound-guided Transversus Abdominis Plane Block After Hysterectomy
Acronym: TAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Irina Gasanova, ASSOC PROFESSOR, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 022010-002
Record Dates: First submitted 2010-06-28; First posted 2010-06-30 (Estimated); Results first posted 2014-04-22 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-01

CONDITIONS: Post Operative Pain
Keywords: Postoperative pain, TAP block, Hysterectomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ketorolac 30 mg, IV + TAP block (Active Comparator): Ketorolac 30 mg, IV + Bilateral ultrasound-guided TAP blocks at the end of the surgery
  First 24-h Postoperative: Ketorolac 30 mg q 6h + acetaminophen 650 mg q6h + IV-PCA morphine
  24-48-h Postoperative: Oral ibuprofen 800 mg q 8 h + hydrocodone/acetaminophen 5mg/500 mg 1-2 tablets q 6h, prn
  Interventions: Procedure: TAP block
- TAP block (Active Comparator): Intraoperative (at the end of surgery): Bilateral ultrasound-guided TAP block at the end of the surgery
  First 24-h Postoperative: IV-PCA morphine
  24-48-h Postoperative: Oral ibuprofen 800 mg q 8 h + hydrocodone/acetaminophen 5mg/500 mg 1-2 tablets q 6h, prn
  Interventions: Procedure: TAP block
- Ketorolac 30 mg (No Intervention): Intraoperative (at the end of surgery): Ketorolac 30 mg, IV at the end of the surgery.
  First 24-h Postoperative: Ketorolac 30 mg q 6h + acetaminophen 650 mg q6h +IV-PCA morphine.
  24-48-h Postoperative: Oral ibuprofen 800 mg q 8 h + hydrocodone/acetaminophen 5mg/500 mg 1-2 tablets q 6h, prn

INTERVENTIONS:
Procedure: TAP block — Group Intraoperative (at the end of surgery): Ketorolac 30 mg, IV + TAP block; TAP block
  First 24-h Postoperative: Ketorolac 30 mg q 6h + acetaminophen 650 mg q6h + IV-PCA morphine
  24-48-h Postoperative: Oral ibuprofen 800 mg q 8 h + hydrocodone/acetaminophen 5mg/500 mg 1-2 tablets q 6h, prn
  Arms: Ketorolac 30 mg, IV + TAP block; TAP block

SUMMARY:
In this randomized, controlled, observer-blinded study we plan to evaluate ultrasound-guided transversus abdominis plane (TAP) block for postoperative pain management in patients undergoing abdominal hysterectomy.

DETAILED DESCRIPTION:
Patients undergoing abdominal hysterectomy (n=75) at Parkland Hospital will be randomized into one of three groups to receive either ultrasound-guided bilateral TAP block with or without NSAIDs and acetaminophen (Groups 1 and 2) or the conventional analgesic regimen (Group 3) for postoperative pain management. The remaining aspect of perioperative care, including the general anesthetic technique, will be standardized and similar for all patients. The duration of the involvement in the study will be until 48 hours postoperatively. The pre-anesthesia care unit personnel will identify patients during their preoperative clinic visit. There will be no incentive or payment to the patients.

Patients in Group 1 and 2 will receive ultrasound-guided bilateral TAP block after surgery. In the first 24-h postoperative period, patients in Groups 1 and 3 will receive acetaminophen 650 mg every 6 h orally, ketorolac 30 mg every 6 h, and morphine via an intravenous patient controlled analgesia (IV-PCA) system to maintain adequate pain control. Patients in Group 2 will receive IV-PCA morphine for the first 24 hours in addition to the ultrasound-guided bilateral block. In the 24-48 h study period, all patients will receive oral ibuprofen 800 mg three times a day and a combination of hydrocodone/acetaminophen 5mg/500 mg 1-2 tablets every 6h, prn. The postoperative analgesia will be documented using the visual analog score (0=no pain,10=worst pain). In addition, total opioid dose over the 48-h study period will be documented. Postoperative nausea will be measured using a categorical scoring system (none=0, mild=1, moderate=2, severe=3) and episodes of vomiting will be documented. Rescue antiemetics will be given to any patient who complains of nausea or vomiting. All variables will be assessed at 2, 6, 12, 24, and 48 hours, postoperatively by an investigator blinded to group allocation.

Primary endpoint will be in about 24 hours after surgery morphine consumption. The secondary endpoints will include the VAS pain score at 6, 12, 24 and 48 hours after surgery and side effects associated with morphine use.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* Female ASA physical status 1-3 scheduled for abdominal hysterectomy
* Able to participate personally or by legal representative in informed consent in English or Spanish

Exclusion Criteria:

* History of relevant drug allergy
* Age less than 18 or greater than 80
* Chronic opioid users who may have a tolerance to opioids
* Psychiatric disturbance
* Inability to understand the study protocol procedures
* Patient refusal

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2010-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irina Gasanova, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UTSW Parkland Health Hospital System, Dallas, Texas, United States

REFERENCES:
- [Derived] Gasanova I, Grant E, Way M, Rosero EB, Joshi GP. Ultrasound-guided transversus abdominal plane block with multimodal analgesia for pain management after total abdominal hysterectomy. Arch Gynecol Obstet. 2013 Jul;288(1):105-11. doi: 10.1007/s00404-012-2698-3. Epub 2013 Jan 6. PMID 23291970

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketorolac 30 mg, IV + TAP Block: Bilateral ultrasound-guided TAP blocks and Ketorolac 30 mg IV at the end of the surgery
  First 24-h Postoperative: Ketorolac 30 mg q 6h + acetaminophen 650 mg q6h and IV-PCA morphine
  24-48-h Postoperative: Oral ibuprofen 800 mg q 8 h + hydrocodone/acetaminophen 5mg/500 mg 1-2 tablets q 6h, prn
- TAP Block: Bilateral ultrasound-guided TAP block at the end of the surgery
  First 24-h Postoperative: IV-PCA morphine
  24-48-h Postoperative: Oral ibuprofen 800 mg q 8 h + hydrocodone/acetaminophen 5mg/500 mg 1-2 tablets q 6h, prn
- Ketorolac 30 mg: Ketorolac 30 mg, IV at the end of surgery
  First 24-h Postoperative: Ketorolac 30 mg q 6h + acetaminophen 650 mg q6h + IV-PCA morphine 24-48-h Postoperative: Oral ibuprofen 800 mg q 8 h + hydrocodone/acetaminophen 5mg/500 mg 1-2 tablets q 6h, prn
Period: Overall Study
Arm/Group | Ketorolac 30 mg, IV + TAP Block | TAP Block | Ketorolac 30 mg
Started | 25 | 25 | 25
Completed | 25 | 24 | 25
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ketorolac 30 mg, IV + TAP Block: Bilateral ultrasound-guided TAP block at the end of the surgery
  First 24-h postoperative: Ketorolac 30 mg, IV, every 6h + acetaminophen 650 mg, orally, every 6h + IV-PCA morphine
- TAP Block: Bilateral ultrasound-guided TAP block at the end of the surgery+ IV-PCA morphine
  First 24-h postoperative: IV-PCA morphine
- Ketorolac 30 mg IV: Ketorolac 30 mg, IV at the end of surgery
  First 24-h postoperative: Ketorolac 30 mg q 6h + acetaminophen 650 mg q6h + IV-PCA morphine
- Total: Total of all reporting groups
Arm/Group | Ketorolac 30 mg, IV + TAP Block | TAP Block | Ketorolac 30 mg IV | Total
Number analyzed (Participants) | 25 | 24 | 25 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (5.4) | 43.8 (6.5) | 43.1 (5.6) | 43.1 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 25 | 74
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 24 | 25 | 74

OUTCOME MEASURES:

1. Primary Outcome: Morphine Consumption
Description: Morphine consumption over the first 24 hours
Time Frame: 24 hours post surgery
Measure: Mean (Standard Deviation); unit: mg
Groups:
- Ketorolac 30 mg: Ketorolac 30 mg after surgery
  First 24-h postoperative: Ketorolac 30 mg q 6h + acetaminophen 650 mg q6h + IV-PCA morphine
Arm/Group | Ketorolac 30 mg, IV + TAP Block | TAP Block | Ketorolac 30 mg
Number analyzed (Participants) | 25 | 24 | 25
mg | 38.4 (25.7) | 38.6 (26.8) | 42.6 (31.2)

ADVERSE EVENTS:
Time Frame: 48-hour study period after surgery
Arm/Group | Ketorolac 30 mg, IV + TAP Block | TAP Block | Ketorolac 30 mg
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/24 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes